CLINICAL TRIAL: NCT02004327
Title: Randomized, Open-label, Single Dose, Crossover Phase I Clinical Study to Evaluate the Pharmacokinetics of DW1029M 300 mg, 600 mg and 1200 mg After Oral Administration in Healthy Male Volunteer
Brief Title: The Phase I Clinical Study to Evaluate the Pharmacokinetics of Dw1029M in Healthy Male Volunteer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong Wha Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DW1029M-I-3
Record Dates: First submitted 2013-11-14; First posted 2013-12-09 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A Group (Experimental): 1. 1st administration - DW1029M300mg PO Once
  2. 2nd administration - DW1029M600mg PO Once
  3. 3rd administration - DW1029M1200mg PO Once
  Interventions: Drug: DW1029M300mg; Drug: DW1029M600mg; Drug: DW1029M1200mg
- B Group (Experimental): 1. 1st administration - DW1029M600mg PO Once
  2. 2nd administration - DW1029M1200mg PO Once
  3. 3rd administration - DW1029M300mg PO Once
  Interventions: Drug: DW1029M300mg; Drug: DW1029M600mg; Drug: DW1029M1200mg
- C Group (Experimental): 1. 1st administration - DW1029M1200mg PO Once
  2. 2nd administration - DW1029M300mg PO Once
  3. 3rd administration - DW1029M600mg PO Once
  Interventions: Drug: DW1029M300mg; Drug: DW1029M600mg; Drug: DW1029M1200mg

INTERVENTIONS:
Drug: DW1029M300mg — DW1029M300mg PO Once
  Other Names: DW1029M300mg 1 tablet
Drug: DW1029M600mg — DW1029M300mg 2 tablets Once
  Other Names: DW1029M300mg 2 tablets
Drug: DW1029M1200mg — DW1029M300mg 4 tablets PO Once
  Other Names: DW1029M300mg 4 tablets

SUMMARY:
1. Objective After single dose in healthy adults the capacity of the Group for DW1029M evaluate the pharmacokinetic characteristics.
2. Indication Diabetic kidney disease
3. Efficacy

   1. Primary

      * AUClast, AUCinf, AUClast/D, AUCinf/D
      * Cmax, Cmax/D
   2. Secondary

      * Tmax, t1/2, CL/F, Vz/F
4. Safety

   1. Adverse Event Monitoring
   2. V/S, EKG, Laboratory Test, P/E

DETAILED DESCRIPTION:
Healthy volunteers for clinical trials targeting drug administration date (1d) within 3 weeks from the (-21d ~-1d) in the interview, physical examination and laboratory tests , including through the screening is performed.

Through screening deems appropriate in this clinical trial is intended for the final subjects randomized to three groups to order .

The first phase one clinical trial subjects performed one day before (the -1 ) 18:00 Chonbuk National University Hospital, convened as a physical examination and perform hwalryeong signs .

One person to dinner , except for the drinking water should be fasting . One clinical trials (the first day) 20:00 subjects randomly assigned to groups according to the order in which the test is administered in a single oral medication .

The subjects for clinical trials with 240 mL water, medicines and swallow whole , chew before swallowing drugs should .

Blood according to the schedule after the clinical trial , including vital signs and physical examination is performed. The subjects that had a fixed schedule and is discharged on the morning of the second .

Is at least one week washout period . Since the two groups according to the order group and three creeping dose , except for the one the same tiles to proceed.

After a period of three clinical trials, three day period from taking drugs for clinical trials after 3-5 days to perform the post-study visit .

ELIGIBILITY:
Inclusion Criteria:

* More than 20 years of age at the time of screening and less than 55 years old healthy male
* (17.5 ~ 30.5 kg/m2 body mass index (BMI) and weight 45 kg or more

  ☞ body mass index (BMI) = weight (kg) / height (m) 2
* No congenital or chronic diseases, internal medicine examination results who does not have psychotic symptoms or findings

Exclusion Criteria:

* Clinically significant blood, kidney, endocrine, respiratory, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but, at the time of administration of seasonal allergic untreated asymptomatic except for sex), medical history or evidence
* Drugs that may affect the absorption of all the states (eg, gastrectomy)
* Investigational drugs within two months before the first dose participated in other clinical trials

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-12; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Maximum Concentration of DW1029M in plasma | 24 hours

SECONDARY OUTCOMES:
Area under concentration-time curve of DW1029M in plasma | 24hours
Time to maximal concentration of DW1029M in Plasma | 24hours
Elimination half time of DW1029M in Plasma | 24hours
Apparent clearance of DW1029M in Plasma | 24hours
Apparent volume of distribution of DW1029M in Plasma | 24hours

CONTACTS AND LOCATIONS:
Overall Officials: Cheol-hee Lim, CR Manager, Study Director — DongWha Pharmaceutical Company
Locations (1):
- Chonbuk National University Hospital, Jeonju-si, Jeollabuk-do, Geonjiro, Deokjin-gu, South Korea